CLINICAL TRIAL: NCT02162498
Title: Effect of Feeding Buddies on Adherence to WHO PMTCT Guidelines in South Africa
Brief Title: Study to Determine Impact of Feeding Buddies on Adherence to WHO PMTCT Guidelines in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: University of KwaZulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD075090-02 (NIH)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-08

CONDITIONS: HIV; PMTCT
Keywords: Peer support; Adherence; Exclusive breastfeeding; Early infant diagnosis; Stigma and disclosure
MeSH Terms: conditions — Breast Feeding; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feeding buddies intervention (Experimental): Sites receiving a comprehensive feeding buddy program implemented by the Window of Opportunity program.
  Interventions: Behavioral: Feeding buddies
- Standard of care (No Intervention): Sites from Window of Opportunity program who are not yet receiving the comprehensive feeding buddies program and are only receiving standard of care PMTCT support.

INTERVENTIONS:
Behavioral: Feeding buddies — The Window of Opportunity program is implementing feeding buddies within their comprehensive programming. Their feeding buddies intervention targets all mothers at ANC for promoting health behaviors, especially exclusive breastfeeding.
  The NIH study is an implementation science award to evaluate the feeding buddies intervention, specifically among HIV positive recipients and evaluating the outcome of adherence to PMTCT recommendations.
  Arms: Feeding buddies intervention

SUMMARY:
The 2010 revised WHO recommendations to provide antiretroviral (ARV) prophylaxis or treatment to mothers or infants during the breastfeeding period indicate a paradigm shift in prevention of mother-to-child transmission (PMTCT); care; and treatment programming. Yet despite South Africa's adoption of this guidance, myriad challenges currently exist. Confusion in the public health care system related to mixed messaging around safe infant feeding and the provision of-and now withdrawal of-free formula milk have made adherence to exclusive breastfeeding a challenge in South Africa. Cultural, social, and psychological factors influence the ability of women to follow PMTCT guidelines, which include exclusive breastfeeding for six months, adherence to ARV prophylaxis or treatment, and early infant diagnosis. Facility-based interventions alone are often inadequate to effect sustained behavioral changes in the face of multiple contextual factors. Community- and home-based support are needed, yet cost and systems constraints make these infeasible in many PMTCT programs. Some preliminary pilot data suggests that a feeding buddy strategy could fill this gap and provide a home-based support system for the mother. The feeding buddy, who is selected by an HIV-positive pregnant woman to support her in overcoming sociocultural challenges to adhering to various aspects of PMTCT programs, is not an employed health care worker, but rather an individual known to the mother, making the intervention extremely cost-effective, and requiring minimal resources to implement. In the Uthungulu District of KZN the Programme for Appropriate Technologies in Health (PATH) is implementing a programme (Window of Opportunity-WinOp) of improving health of mothers and infants, and the feeding buddy strategy is one of the strategies included in this overall package of care. While this strategy has been encouraged by the South African Department of Health, it has not previously been implemented nor obviously evaluated. In order to scale-up such a programme and justify the human resource costs, it is vital that such a programme be evaluated.

The goal of this proposed research study is therefore to evaluate the effect of the feeding buddy strategy to support mothers to adhere to PMTCT recommendations.

The investigators hypothesize that mothers who choose a feeding buddy will have increased rates of exclusive breastfeeding and adherence to ARV prophylaxis or treatment, as well as improved rates of early infant diagnosis and stigma reduction.

This evaluation will provide valuable information to the Department of Health in terms of choosing best practice models for promoting HIV-free infant survival and optimum health of infants in resource limited settings. The project plans to employ a cluster randomized intervention design and will include 300 mothers and their infants as well as the 300 buddies in the intervention group, as well as 300 mothers in the control group. All participants will be part of the WinOp feeding buddy intervention programme.

ELIGIBILITY:
Inclusion criteria for pregnant women

* Pregnant women 18 years of age or older and attending one of the study clinics and enrolled in the national PMTCT program
* Women must be least 14 but not more than 28 weeks pregnant (defined using the date of the last menstrual period and clinical examination)
* They must have a documented HIV infection
* Have indicated their intention to deliver and remain within the study area for at least 6 months following the birth of their infant
* Committed to exclusively breastfeed
* Provide written informed consent
* Intervention mothers only: Must have agreed to participate in the WinOp feeding buddies program, and identified and disclosed to a feeding buddy

Exclusion criteria for pregnant women

* Women will be excluded from the study if they do not attend a study clinic
* If they are more than 28 weeks pregnant before enrollment
* If they indicate their intention to deliver or have postnatal visits outside the study area
* Intend to formula or mixed feed their infant
* Any participant that is seriously ill will be excluded from the study and referred for services and support
* Intervention mothers only: Not participating in the WinOp feeding buddies program

Inclusion criteria for buddies

* Participants will include people of any gender who are 18 years of age or older, who the mother has selected - HIV status will not be an inclusion criteria for this feeding buddy.
* Provide written informed consent

Exclusion criteria for buddies

* Potential participants will be excluded who are under the age of 18. HIV status is not an exclusion criteria for the feeding buddy.
* Any participant that is seriously ill will be excluded from the study and referred for services and support

Inclusion criteria for community care givers and PMTCT counselors (in-depth interviews only)

* Participants will include people of any gender who are 18 years of age or older, who serve as a community care giver or PMTCT counselor in the study sites.
* Provide written informed consent

Exclusion criteria for community care givers and PMTCT counselors (in-depth interviews only)

* Potential participants will be excluded who are under the age of 18 and who do not serve as a community care giver or PMTCT counselor in a study site.
* Any participant that is seriously ill will be excluded from the study and referred for services and support

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 932 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To determine the effect of a feeding buddy on adherence to exclusive breastfeeding. | 6 months postpartum
  We hypothesize that mothers who choose a feeding buddy to provide enhanced support will have increased rates of initiation and duration of exclusive breastfeeding.
  Exclusive breastfeeding: Defined as no other food or drink, not even water, apart from breast milk (including expressed breast milk) with the exception of drops or syrups consisting of vitamins, mineral supplements or medicines (WHO/UNICEF. Infant and young child feeding counselling: an integrated course. Geneva: World Health Organization; 2006), measured by recall prior to each visit; from this aggregate data number of months engaged in EBF will be calculated.
To determine the effect of a feeding buddy on adherence to ARV prophylaxis or ART regimens. | 6 months postpartum
  We hypothesize that mothers who choose a feeding buddy to provide enhanced support will have increased rates of adherence to ARV prophylaxis or ART regimens.
  Adherence to ARV: Three separate outcomes will be examined, including adherence to:
  1. ARV prophylaxis to prevent MTCT among HIV+ mothers who do not have indications for ARV treatment
  2. ARV treatment of HIV+ mothers when indicated for their own health
  3. ARV prophylaxis of infant
  Adherence to ARV in each case defined as taking more than 95% of prescribed doses.71 Adherence will be assessed through:
  1. Medical records at each clinic visit (e.g., pill counts) &
  2. Self-report at study visits Dose adherence is measured as number of prescribed doses per drug per day divided by the self-reported number of missed doses on each of the past four days. In addition, an adherence index 71 is based on dosing, timing and special instructions questions.

SECONDARY OUTCOMES:
To determine the effect of a feeding buddy on adherence to infant HIV testing at 6 weeks. | 6 weeks postpartum
  We hypothesize that mothers who choose a feeding buddy to provide enhanced support will have increased rates of having their infant tested for HIV at 6 weeks.
  Early infant HIV diagnosis: This will be examined through date of infant HIV PCR test as indicated through recall and medical record.
To determine the effect of a feeding buddy on disclosure and stigma. | 6 months postpartum
  We hypothesize that mothers who choose a feeding buddy will have increased rates of disclosure and decreased effect from stigma around HIV status.
  Impact on stigma and disclosure: This will be measured through descriptive analysis of perceived and enacted stigma associated with being HIV.
  Exposure: The exposure of interest is choosing a feeding buddy and level of exposure to the feeding buddy, the latter providing a dose-response measure of support. Exposure will be measured as having selected a buddy who has attended an orientation session (yes/no); number of visits to antenatal and postnatal visits accompanied by the feeding buddy; and the number, frequency, and type (in-person, telephone) of contacts between mother and buddy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of KwaZulu-Natal, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Gavine A, Shinwell SC, Buchanan P, Farre A, Wade A, Lynn F, Marshall J, Cumming SE, Dare S, McFadden A. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2022 Oct 25;10(10):CD001141. doi: 10.1002/14651858.CD001141.pub6. PMID 36282618